CLINICAL TRIAL: NCT04374123
Title: COVID-19 Serologic Screening and a Strict Protocol in the Management of a Referral Gastrointestinal Endoscopy Unit: a Prospective Study
Brief Title: COVID-19 Serology Screening and Strict Protocol in the Endoscopy Unit
Status: Completed | Type: Observational
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Sponsor
Other Study IDs: IECED-04-15-covid
Record Dates: First submitted 2020-04-20; First posted 2020-05-05 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: COVID

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Serological screening for IgG and IgM antibodies against COVID-19 — Serum evaluation for IgG and IgM antibodies against COVID-19 in patients in the endoscopy unit during the COVID 19 pandemic

SUMMARY:
The novel COronaVIrus Disease 19 (COVID-19) outbreak has impacted daily activities in nearly 210 countries and territories worldwide. In Ecuador, the city of Guayaquil has nearly two-thirds of the COVID-positive patients in the country and nearly 40% of infected individuals are health-care related personnel.

Nonemergent, emergent and urgent endoscopic procedures are necessary to be performed during the COVID-19 pandemic. Several experiences in the management of the endoscopic unit during the pandemic has been proposed. We aimed to prospectively evaluate a strict protocol for preventing potential nosocomial infection of COVID-19.

DETAILED DESCRIPTION:
Consecutive patients with appointment for endoscopic examination and procedures will be contacted via a telephone call by a pulmonologist, who will perform a triage with a screening questionnaire between 24-48 hours before the scheduled procedure. The pulmonologist will seek for history of fever, respiratory symptoms, and/or close-contacts COVID-patients. After exclusion of all respiratory symptoms or history suggestive of COVID-19, patients will be evaluated for serum IgG and IgM levels using a rapid test.

Only after complete evaluation and revision of serological levels, body temperature will be measure before entering the endoscopy unit. Patients will be isolated in an individual preoperative and recovery room after the endoscopic procedure, avoiding contacts with other patients. The endoscopy staff (endoscopists, nurses, administrative personal, anesthesia staff) will use personal protective equipment (PPE) including N95 face mask, face shield, shoe covers, gowns, and gloves.

All the staff will be evaluated for nucleic acid PCR testing within three days before resuming activities in the endoscopy unit, all staff members will be evaluated for respiratory symptoms and changes in body temperature before starting daily activities. At the end of the study all the staff will be evaluated for IgM and IgG antibodies against COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to participate
* Available serum samples for IgG and IgG antibodies against COVID-19
* Ability to complete the screening questionnaire

Exclusion Criteria:

* Patients with respiratory symptoms
* Patients with COVID-19 active infection

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients from the Endoscopy Unit at the Instituto Ecuatoriano de Enfermedades Digestivas, Guayaquil, Ecuador. Patients that completed screening questionnaire and serological screening for COVID-109 before the performance of the endoscopic procedures.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Rate of COVID-19 nosocomial infection among the endoscopy staff at the end of the 30-days study. | through study completion, an average of 30 days
  COVID-19 infection in the staff documented via PCR
Numbers of patients evaluated and treated during the COVID-19 outbreak in the endoscopy unit at the end of the 30-days study. | through study completion, an average 30 days
  Endoscopic records of patients treated during the COVID-19 protocol
Technical success rate of endoscopic procedures during the 30-days study period. | through study completion, an average 30 days
  technical success of endoscopic procedures
IgG and IgM against COVID-19 in the endoscopy staff measured at the end of the study. | through study completion, an average 30 days
  serum levels of IgG and IgM against COVID-19
Adverse events rate of endoscopic procedures during the 30-days | through study completion, an average 30 days
  adverse events of endoscopic procedures

CONTACTS AND LOCATIONS:
Locations (1):
- Ecuadorian Institute of Digestive Diseases, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Han J, Wang Y, Zhu L, Cui Y, Li L, Zeng Z, Zhang S. Preventing the spread of COVID-19 in digestive endoscopy during the resuming period: meticulous execution of screening procedures. Gastrointest Endosc. 2020 Aug;92(2):445-447. doi: 10.1016/j.gie.2020.03.3855. Epub 2020 Apr 5. No abstract available. PMID 32268134
- [Result] Repici A, Pace F, Gabbiadini R, Colombo M, Hassan C, Dinelli M; ITALIAN GI-COVID19 Working Group. Endoscopy Units and the Coronavirus Disease 2019 Outbreak: A Multicenter Experience From Italy. Gastroenterology. 2020 Jul;159(1):363-366.e3. doi: 10.1053/j.gastro.2020.04.003. Epub 2020 Apr 10. No abstract available. PMID 32283102
- [Result] Thompson CC, Shen L, Lee LS. COVID-19 in endoscopy: Time to do more? Gastrointest Endosc. 2020 Aug;92(2):435-439. doi: 10.1016/j.gie.2020.03.3848. Epub 2020 Mar 29. No abstract available. PMID 32234312